CLINICAL TRIAL: NCT03794284
Title: Performance of a Multiplex PCR -Microarray-based Assay in the Detection of Mycobacterium Tuberculosis and Non-tuberculous Mycobacterium Species in Smear-positive Pulmonary Clinical Specimens
Brief Title: Multiplex PCR -Microarray-based Assay in the Detection of Mycobacterium
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Assistant Professor and Head, Division of Infectious Diseases, Chinese University of Hong Kong
Other Study IDs: VereMTB_v2_24_10_2018
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Tuberculosis; Non-Tuberculous Mycobacterial Pneumonia
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At least 2mL of sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: VereMTB — At least 2 mL of patient's expectorated or induced sputum would be collected for VereMTB assay and their clinical data would be retrieved for analysis use.

SUMMARY:
The study will use the VereMTB tool for rapid diagnosis of TB or non-tuberculous mycobacterium (NTM) pulmonary infections in hospitalised patients, with positive results in acid-fast bacilli smears, which are emerging in many regions of the world.

DETAILED DESCRIPTION:
Delay in diagnosis and treatment of tuberculosis was common in hospitalised patients all around the world, and was associated with poorer outcomes, including respiratory failure and mortality. Rapid and accurate tools for diagnosis of TB is of great importance in initial treatment and for better treatment outcomes. Other than TB, non-tuberculous mycobacterium (NTM) pulmonary infections are emerging in many regions of the world. These bacterium are more common to be found in respiratory specimens than MTB. With similar clinical presentation of NTM pulmonary infections and pulmonary TB, misdiagnosis of NTM pulmonary infections to pulmonary TB would lead to unnecessary intake of anti-TB medications and delay of the initiation of corresponding treatment.

This test aims to detect MTB as well differentiate the NTM species involved in pulmonary infections simultaneously using VereMTB.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. One or more symptoms compatible with mycobacterial pulmonary infections, including fever, cough, sputum production,hemoptysis dyspnea, chest pain and weight loss
3. One or more sputum samples with positive AFB smear

Exclusion Criteria:

1. Receiving anti-mycobacterial treatment for more than one week
2. Refusal to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Prince of Wales Hospital with suspected pulmonary TB with positive AFB smears will be identified by Infectious Diseases physicians and recruited accordingly.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
diagnostic test correlation | 6 months from the date of first recruitment
  Sensitivity, specificity, positive predictive value, and negative predictive value, will be calculated to determine accuracy of VereMTB, in diagnosing MTB and NTM

CONTACTS AND LOCATIONS:
Overall Officials: Chung Yan Grace Lui, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD Tuberculosis Collaborators. The global burden of tuberculosis: results from the Global Burden of Disease Study 2015. Lancet Infect Dis. 2018 Mar;18(3):261-284. doi: 10.1016/S1473-3099(17)30703-X. Epub 2017 Dec 7. PMID 29223583
- [Background] Lui G, Wong RY, Li F, Lee MK, Lai RW, Li TC, Kam JK, Lee N. High mortality in adults hospitalized for active tuberculosis in a low HIV prevalence setting. PLoS One. 2014 Mar 18;9(3):e92077. doi: 10.1371/journal.pone.0092077. eCollection 2014. PMID 24642794
- [Background] Bhurayanontachai R, Maneenil K. Factors influencing development and mortality of acute respiratory failure in hospitalized patient with active pulmonary tuberculosis: a 10-year retrospective review. J Thorac Dis. 2016 Jul;8(7):1721-30. doi: 10.21037/jtd.2016.06.22. PMID 27499962
- [Background] Namkoong H, Kurashima A, Morimoto K, Hoshino Y, Hasegawa N, Ato M, Mitarai S. Epidemiology of Pulmonary Nontuberculous Mycobacterial Disease, Japan. Emerg Infect Dis. 2016 Jun;22(6):1116-7. doi: 10.3201/eid2206.151086. No abstract available. PMID 27191735
- [Background] Kim HS, Lee Y, Lee S, Kim YA, Sun YK. Recent trends in clinically significant nontuberculous Mycobacteria isolates at a Korean general hospital. Ann Lab Med. 2014 Jan;34(1):56-9. doi: 10.3343/alm.2014.34.1.56. Epub 2013 Dec 6. PMID 24422197
- [Background] Chien JY, Lai CC, Sheng WH, Yu CJ, Hsueh PR. Pulmonary infection and colonization with nontuberculous mycobacteria, Taiwan, 2000-2012. Emerg Infect Dis. 2014 Aug;20(8):1382-5. doi: 10.3201/eid2008.131673. PMID 25062534
- [Background] Lan R, Yang C, Lan L, Ou J, Qiao K, Liu F, Gao Q. Mycobacterium tuberculosis and non-tuberculous mycobacteria isolates from HIV-infected patients in Guangxi, China. Int J Tuberc Lung Dis. 2011 Dec;15(12):1669-75. doi: 10.5588/ijtld.11.0036. PMID 22118176
- [Background] McCarthy KD, Cain KP, Winthrop KL, Udomsantisuk N, Lan NT, Sar B, Kimerling ME, Kanara N, Lynen L, Monkongdee P, Tasaneeyapan T, Varma JK. Nontuberculous mycobacterial disease in patients with HIV in Southeast Asia. Am J Respir Crit Care Med. 2012 May 1;185(9):981-8. doi: 10.1164/rccm.201107-1327OC. Epub 2012 Feb 16. PMID 22345581
- [Background] Cabibbe AM, Miotto P, Moure R, Alcaide F, Feuerriegel S, Pozzi G, Nikolayevskyy V, Drobniewski F, Niemann S, Reither K, Cirillo DM; TM-REST Consortium; TB-CHILD Consortium. Lab-on-Chip-Based Platform for Fast Molecular Diagnosis of Multidrug-Resistant Tuberculosis. J Clin Microbiol. 2015 Dec;53(12):3876-80. doi: 10.1128/JCM.01824-15. Epub 2015 Aug 5. PMID 26246486
- [Background] Lazzeri E, Santoro F, Oggioni MR, Iannelli F, Pozzi G. Novel primer-probe sets for detection and identification of mycobacteria by PCR-microarray assay. J Clin Microbiol. 2012 Nov;50(11):3777-9. doi: 10.1128/JCM.02300-12. Epub 2012 Sep 12. PMID 22972818
- [Background] Hoefsloot W, van Ingen J, Andrejak C, Angeby K, Bauriaud R, Bemer P, Beylis N, Boeree MJ, Cacho J, Chihota V, Chimara E, Churchyard G, Cias R, Daza R, Daley CL, Dekhuijzen PN, Domingo D, Drobniewski F, Esteban J, Fauville-Dufaux M, Folkvardsen DB, Gibbons N, Gomez-Mampaso E, Gonzalez R, Hoffmann H, Hsueh PR, Indra A, Jagielski T, Jamieson F, Jankovic M, Jong E, Keane J, Koh WJ, Lange B, Leao S, Macedo R, Mannsaker T, Marras TK, Maugein J, Milburn HJ, Mlinko T, Morcillo N, Morimoto K, Papaventsis D, Palenque E, Paez-Pena M, Piersimoni C, Polanova M, Rastogi N, Richter E, Ruiz-Serrano MJ, Silva A, da Silva MP, Simsek H, van Soolingen D, Szabo N, Thomson R, Tortola Fernandez T, Tortoli E, Totten SE, Tyrrell G, Vasankari T, Villar M, Walkiewicz R, Winthrop KL, Wagner D; Nontuberculous Mycobacteria Network European Trials Group. The geographic diversity of nontuberculous mycobacteria isolated from pulmonary samples: an NTM-NET collaborative study. Eur Respir J. 2013 Dec;42(6):1604-13. doi: 10.1183/09031936.00149212. Epub 2013 Apr 18. PMID 23598956